CLINICAL TRIAL: NCT02324673
Title: A Phase 1/2 Study to Assess the Pharmacokinetics and Safety of Multiple Doses of Pharmaceutical Cannabidiol Oral Solution in Pediatric Participants With Treatment-Resistant Seizure Disorders
Brief Title: Cannabidiol Oral Solution in Pediatric Participants With Treatment-resistant Seizure Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INS011-14-029
Record Dates: First submitted 2014-12-12; First posted 2014-12-24 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Seizures
Keywords: Treatment-resistant seizures
MeSH Terms: conditions — Seizures | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose Cannabidiol Oral Solution [10 mg/kg/day] (Experimental): Low Dose [10 milligrams/kilogram/day (mg/kg/day)] oral solution containing pharmaceutical grade cannabidiol (nonplant-based). Starting dose of 5 mg/kg in the morning on Day 1 followed by total dose of 10 mg/kg/day (5 mg/kg in the morning and 5 mg/kg in the evening) on Days 4 to 10.
  Interventions: Drug: Cannabidiol Oral Solution
- Mid Dose Cannabidiol Oral Solution [20 mg/kg/day] (Experimental): Mid Dose [20 mg/kg/day] oral solution containing pharmaceutical grade cannabidiol (nonplant-based). Starting dose of 10 mg/kg in the morning on Day 1 followed by total dose of 20 mg/kg/day (10 mg/kg in the morning and 10 mg/kg in the evening) on Days 4 to 10.
  Interventions: Drug: Cannabidiol Oral Solution
- High Dose Cannabidiol Oral Solution [40 mg/kg/day] (Experimental): High Dose [40 mg/kg/day] oral solution containing pharmaceutical grade cannabidiol (nonplant-based). Starting dose of 20 mg/kg in the morning on Day 1 followed by total dose of 40 mg/kg/day (20 mg/kg in the morning and 20 mg/kg in the evening) on Days 4 to 10.
  Interventions: Drug: Cannabidiol Oral Solution

INTERVENTIONS:
Drug: Cannabidiol Oral Solution — An oral solution containing pharmaceutical grade cannabidiol (nonplant-based).

SUMMARY:
This is a Phase 1/2, open-label trial designed to assess the pharmacokinetics, safety, tolerability, and preliminary efficacy of 3 multiple ascending doses of Cannabidiol Oral Solution in a sequential fashion.

Participants will be pediatric (aged 1-17, inclusive), experiencing treatment-resistant seizures, and satisfy all inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception, including treatment-resistant seizure disorder
* Is able to speak and understand the language in which the study is being conducted, is able to understand the procedures and study requirements and has voluntarily signed and dated an informed consent form approved by the Institutional Review Board before the conduct of any study procedure
* In the opinion of the Investigator, the participants and parent(s)/caregiver(s) are willing and able to comply with the study procedures and visit schedules, including venipuncture, inpatient stay at the study center, dosing at the study center twice a day as needed while an outpatient), and the Follow-up Visits (if applicable)

Exclusion Criteria:

* Participant or parent(s)/caregiver(s) have daily commitments during the study duration that would interfere with attending all study visits
* History or current use of dietary supplements, drugs or over-the counter medications outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2016-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Parikh, Study Director — INSYS Therapeutics Inc
Locations (10):
- United States (10):
  - University of California San Francisco Medical Center, San Francisco, California
  - Miami Children's Hospital, Miami, Florida
  - Child Neurology Center - NW F, Pensacola, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Clinical Research Center of Nevada LLC, Las Vegas, Nevada
  - Oregon Health Services University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Texas Scottish Rite Hospital for Children, Dallas, Texas
  - Mary Bridge Children's Hospital, Tacoma, Washington

REFERENCES:
- [Derived] Wheless JW, Dlugos D, Miller I, Oh DA, Parikh N, Phillips S, Renfroe JB, Roberts CM, Saeed I, Sparagana SP, Yu J, Cilio MR; INS011-14-029 Study Investigators. Pharmacokinetics and Tolerability of Multiple Doses of Pharmaceutical-Grade Synthetic Cannabidiol in Pediatric Patients with Treatment-Resistant Epilepsy. CNS Drugs. 2019 Jun;33(6):593-604. doi: 10.1007/s40263-019-00624-4. PMID 31049885

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Started | 20 | 20 | 21
Completed | 20 | 20 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population (SAF), all participants who received ≥1 dose of the investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day] | Total
Number analyzed (Participants) | 20 | 20 | 21 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (5.32) | 7.7 (5.17) | 7.8 (5.39) | 7.6 (5.21)
Age, Customized [Count of Participants; unit: Participants]
  Infants = 1 to <2 years | 5 | 5 | 5 | 15
  Children = 2 to <12 years | 9 | 9 | 10 | 28
  Adolescents = 12 to ≤17 years | 6 | 6 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 11 | 28
  Male | 10 | 13 | 10 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 21 | 61

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for Cannabidiol and Metabolite 7-hydroxy (7-OH) Cannabidiol
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2 years: Day 1 at 2, 4, 8, 12 hours post-dose; Participants ages 2 to <6 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24 and 48 hours post-dose; Participants ages 6 to ≤17 years: Day 1 pre-dose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose.
Time Frame: Day 1 at age-specific times
Population: Pharmacokinetic population (PK), all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for Cmax.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
nanograms/milliliter (ng/mL)
  Cannabidiol | 59.03 (99.98) | 110.5 (142.3) | 256.9 (351.9)
  7-OH Cannabidiol | 28.71 (26.72) | 61.89 (72.88) | 140.9 (210.0)

2. Primary Outcome: Cmax for Cannabidiol and Metabolite 7-OH Cannabidiol
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2 years: Day 10 pre-dose and at 2, 4, 8 and 12 hours post-dose; Participants ages 2 to <6 years: Day 10 pre-dose and at 1, 2, 3, 4, 8, 12 and 24 hours post-dose; Participants ages 6 to ≤17 years: Day 10 pre-dose and at 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
Time Frame: Day 10 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ng/mL
  Cannabidiol: number analyzed (Participants) | 20 | 17 | 21
  Cannabidiol | 119.6 (105.0) | 220.0 (294.7) | 426.8 (327.7)
  7-OH Cannabidiol: number analyzed (Participants) | 20 | 17 | 21
  7-OH Cannabidiol | 79.38 (40.82) | 136.6 (140.9) | 286.1 (201.9)

3. Primary Outcome: Dose Normalized Cmax (Cmax/D) for Cannabidiol and Metabolite 7-OH Cannabidiol
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2: Day 1 at 2, 4, 8, 12 hours post-dose; Participants ages 2 to <6: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24 and 48 hours post-dose; Participants ages 6 to ≤17: Day 1 pre-dose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose.
Time Frame: Day 1 at age-specific times
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL/(mg/kg)
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ng/mL/(mg/kg)
  Cannabidiol | 11.72 (19.89) | 10.77 (13.97) | 13.25 (18.07)
  7-OH Cannabidiol | 5.737 (5.330) | 5.990 (7.011) | 7.286 (10.91)

4. Primary Outcome: Cmax/D for Cannabidiol and Metabolite 7-OH Cannabidiol
Description: as for outcome 2
Time Frame: Day 10 at age-specific times
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL/(mg/kg)
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ng/mL/(mg/kg)
  Cannabidiol: number analyzed (Participants) | 20 | 17 | 21
  Cannabidiol | 23.79 (20.46) | 21.16 (28.40) | 21.40 (16.38)
  7-OH Cannabidiol: number analyzed (Participants) | 20 | 17 | 21
  7-OH Cannabidiol | 15.82 (7.928) | 13.10 (13.06) | 14.39 (10.26)

5. Primary Outcome: Time to Cmax (Tmax) for Cannabidiol and Metabolite 7-OH Cannabidiol
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2 years: Day 1 at 2, 4, 8, 12 hours post-dose; Participants ages 2 to <6 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24 and 48 hours post-dose; Participants ages 6 to ≤17 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24, 36, 48 and 72 hours post-dose.
Time Frame: Day 1 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for tmax.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
hours (h)
  Cannabidiol | 2.58 [1.02 to 8.00] | 4.00 [1.00 to 8.08] | 3.15 [1.00 to 24.02]
  7-OH Cannabidiol | 2.55 [1.00 to 6.08] | 4.00 [1.00 to 11.95] | 3.07 [1.00 to 12.05]

6. Primary Outcome: Time to Cmax (Tmax) for Cannabidiol and Metabolite 7-OH Cannabidiol
Description: as for outcome 2
Time Frame: Day 10 at age-specific times
Population: as for outcome 5
Measure: Median (Full Range); unit: h
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
h
  Cannabidiol: number analyzed (Participants) | 20 | 17 | 21
  Cannabidiol | 2.99 [1.00 to 4.25] | 2.00 [0.00 to 6.00] | 3.00 [0.00 to 6.02]
  7-OH Cannabidiol: number analyzed (Participants) | 20 | 17 | 21
  7-OH Cannabidiol | 2.08 [1.00 to 4.08] | 2.03 [1.00 to 6.05] | 2.03 [0.00 to 5.90]

7. Primary Outcome: Half Life (t1/2) for Cannabidiol and Metabolite 7-OH Cannabidiol for Participants ≥2 Years of Age
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 2 to <6 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24 and 48 hours post-dose; Participants ages 6 to ≤17 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24, 36, 48 and 72 hours post-dose; Participants ages 1 to <2 years were not included in this analysis.
Time Frame: Day 1 at age-specific times
Population: Participants ≥2 years from the PK Population who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for t1/2.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 15 | 15 | 16
h
  Cannabidiol: number analyzed (Participants) | 11 | 8 | 12
  Cannabidiol | 31.31 (23.46) | 33.48 (14.97) | 21.58 (10.50)
  7-OH Cannabidiol: number analyzed (Participants) | 15 | 13 | 13
  7-OH Cannabidiol | 19.71 (7.640) | 31.84 (24.28) | 14.77 (4.354)

8. Primary Outcome: Elimination Rate (Lambda-z [λz]) for Cannabidiol and Metabolite 7-OH Cannabidiol for Participants ≥2 Years of Age
Description: as for outcome 7
Time Frame: Day 1 at age-specific times
Population: Participants ≥2 years from the PK Population who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for λz.
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 15 | 15 | 16
1/h
  Cannabidiol: number analyzed (Participants) | 11 | 8 | 12
  Cannabidiol | 0.02969 (0.01386) | 0.02836 (0.02340) | 0.03949 (0.01976)
  7-OH Cannabidiol: number analyzed (Participants) | 15 | 13 | 13
  7-OH Cannabidiol | 0.04053 (0.01557) | 0.03276 (0.01985) | 0.05123 (0.01711)

9. Primary Outcome: Oral Clearance (CL/F) for Cannabidiol for Participants ≥2 Years of Age
Description: as for outcome 7
Time Frame: Day 1 at age-specific times
Population: Participants ≥2 years from the PK Population who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for CL/F.
Measure: Mean (Standard Deviation); unit: Liters (L)/h/kg
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 10 | 8 | 12
Liters (L)/h/kg | 29.78 (15.96) | 21.10 (23.04) | 31.29 (30.43)

10. Primary Outcome: Volume of Distribution (Vz/F) of Cannabidiol for Participants ≥2 Years of Age
Description: as for outcome 7
Time Frame: Day 1 at age-specific times
Population: Participants ≥2 years from the PK Population who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for Vz/F.
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 10 | 8 | 12
L/kg | 1021 (609.1) | 930.8 (1034) | 982.6 (1119)

11. Primary Outcome: Area Under the Plasma-Concentration Time Curve From 0 to 12 Hours Post-dose [AUC(0-12)] for Cannabidiol and Metabolite 7-OH Cannabidiol on Day 1
Description: as for outcome 5
Time Frame: Day 1 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for AUC(0-12).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ng*h/mL
  Cannabidiol: number analyzed (Participants) | 20 | 19 | 21
  Cannabidiol | 173.9 (179.6) | 507.1 (687.7) | 914.5 (1155)
  7-OH Cannabidiol: number analyzed (Participants) | 20 | 19 | 21
  7-OH Cannabidiol | 124.4 (80.18) | 329.8 (402.9) | 646.7 (886.3)

12. Primary Outcome: Dose Normalized AUC(0-12) [AUC (0-12)/D] for Cannabidiol and Metabolite 7-OH Cannabidiol on Day 1
Description: as for outcome 5
Time Frame: Day 1 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for AUC(0-12)/D.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ng*h/mL
  Cannabidiol: number analyzed (Participants) | 20 | 19 | 21
  Cannabidiol | 34.60 (35.48) | 49.23 (66.68) | 47.13 (59.38)
  7-OH Cannabidiol: number analyzed (Participants) | 20 | 19 | 21
  7-OH Cannabidiol | 24.88 (15.93) | 31.77 (38.00) | 33.39 (45.94)

13. Primary Outcome: AUC From Time 0 to the Last Quantifiable Concentration [AUC(0-last)] on Day 1 for Cannabidiol and Metabolite 7-OH Cannabidiol on Day 1 for Participants ≥2 Years of Age
Description: as for outcome 7
Time Frame: Day 1 at age-specific times
Population: Participants ≥2 years from the PK Population who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for AUC(0-last).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 15 | 15 | 16
ng*h/mL
  Cannabidiol | 250.0 (217.1) | 692.5 (826.9) | 1355 (1447)
  7-OH Cannabidiol | 212.2 (112.1) | 544.9 (526.6) | 1221 (1296)

14. Primary Outcome: AUC From Time 0 to Infinity [AUC(0-inf)] for Cannabidiol and Metabolite 7-OH Cannabidiol on Day 1 for Participants ≥2 Years of Age
Description: as for outcome 7
Time Frame: Day 1 at age-specific times
Population: Participants ≥2 years from the PK Population who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for AUC(0-inf).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 15 | 15 | 16
ng*h/mL
  Cannabidiol: number analyzed (Participants) | 10 | 8 | 12
  Cannabidiol | 270.1 (256.7) | 1140 (1118) | 1584 (1709)
  7-OH Cannabidiol: number analyzed (Participants) | 15 | 11 | 13
  7-OH Cannabidiol | 229.3 (122.3) | 704.1 (627.8) | 1354 (1428)

15. Primary Outcome: Dose Normalized AUC(0-inf) [AUC(0-inf)/D] for Cannabidiol and Metabolite 7-OH Cannabidiol on Day 1 for Participants ≥2 Years of Age
Description: as for outcome 7
Time Frame: Day 1 at age-specific times
Population: Participants ≥2 years from the PK Population who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for AUC(0-inf)/D.
Measure: Mean (Standard Deviation); unit: ng*h/mL/(mg/kg)
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 15 | 15 | 16
ng*h/mL/(mg/kg)
  Cannabidiol: number analyzed (Participants) | 10 | 8 | 12
  Cannabidiol | 53.64 (50.04) | 111.8 (111.2) | 83.10 (87.93)
  7-OH Cannabidiol: number analyzed (Participants) | 15 | 11 | 13
  7-OH Cannabidiol | 46.07 (24.63) | 68.43 (62.34) | 70.34 (73.66)

16. Primary Outcome: Metabolite (7-OH Cannabidiol) to Parent (Cannabidiol) Ratio for Cmax [MRCmax] on Day 1
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2 years: Day 1 at 2, 4, 8, 12 hours post-dose; Participants ages 2 to <6 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24 and 48 hours post-dose; Participants ages 6 to ≤17 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24, 36, 48 and 72 hours post-dose.
  MRCmax was adjusted for molecular weight differences between cannabidiol (341.46) and 7-OH cannabidiol (330.46).
Time Frame: Day 1 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for MRCmax.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ratio | 0.8935 (0.5543) | 0.9328 (0.8332) | 0.8081 (0.4849)

17. Primary Outcome: MRCmax on Day 10
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2 years: Day 10 pre-dose and at 2, 4, 8 and 12 hours post-dose; Participants ages 2 to <6 years: Day 10 pre-dose and at 1, 2, 3, 4, 8, 12 and 24 hours post-dose; Participants ages 6 to ≤17 years: Day 10 pre-dose and at 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
  MRCmax was adjusted for molecular weight differences between cannabidiol (341.46) and 7-OH cannabidiol (330.46).
Time Frame: Day 10 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for metabolite to parent ratio.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 17 | 21
ratio | 0.7717 (0.3960) | 0.8230 (0.3880) | 0.7657 (0.4179)

18. Primary Outcome: Metabolite to Parent Ratio for AUC(0-inf) [MRAUC(0-inf)] on Day 1 for Participants ≥2 Years of Age
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 2 to <6 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24 and 48 hours post-dose; Participants ages 6 to ≤17 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24, 36, 48 and 72 hours post-dose; Participants ages 1 to <2 years were not included in this analysis.
  MRAUC(0-inf) was adjusted for molecular weight differences between cannabidiol (341.46) and 7-OH cannabidiol (330.46).
Time Frame: Day 1 at age-specific times
Population: Participants ≥2 years from the PK Population who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for MRAUC(0-inf).
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 10 | 8 | 12
ratio | 0.9099 (0.5173) | 0.9459 (0.4874) | 0.9538 (0.4370)

19. Primary Outcome: Metabolite to Parent Ratio for AUC(0-12) [MRAUC(0-12)] on Day 1
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2 years: Day 1 at 2, 4, 8, 12 hours post-dose; Participants ages 2 to <6 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24 and 48 hours post-dose; Participants ages 6 to ≤17 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24, 36, 48 and 72 hours post-dose.
  MRAUC(0-12) was adjusted for molecular weight differences between cannabidiol (341.46) and 7-OH cannabidiol (330.46).
Time Frame: Day 1 at age-specific times
Population: Participants ≥2 years from the PK Population who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for MRAUC(0-12).
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 19 | 21
ratio | 0.9309 (0.5229) | 0.9793 (0.7147) | 0.9085 (0.5075)

20. Primary Outcome: Metabolite to Parent Ratio for AUC(0-12) [MRAUC(0-12)] on Day 10
Description: Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2 years: Day 10 pre-dose and at 2, 4, 8 and 12 hours post-dose; Participants ages 2 to <6 years: Day 10 pre-dose and at 1, 2, 3, 4, 8, 12 and 24 hours post-dose; Participants ages 6 to ≤17 years: Day 10 pre-dose and at 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
  MRAUC(0-12) was adjusted for molecular weight differences between cannabidiol (341.46) and 7-OH cannabidiol (330.46).
Time Frame: Day 10 at age-specific times
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 19 | 17 | 21
ratio | 0.8795 (0.4084) | 0.7866 (0.2361) | 0.8700 (0.4304)

21. Primary Outcome: AUC(0-12) for Cannabidiol and Metabolite 7-OH Cannabidiol on Day 10
Description: as for outcome 2
Time Frame: Day 10 at age-specific times
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ng*h/mL
  Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  Cannabidiol | 581.6 (283.4) | 1098 (976.4) | 2708 (1789)
  7-OH Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  7-OH Cannabidiol | 513.4 (269.0) | 832.8 (675.2) | 2165 (1405)

22. Primary Outcome: Dose Normalized AUC(0-12) [AUC (0-12)/D] for Cannabidiol and Metabolite 7-OH Cannabidiol on Day 10
Description: as for outcome 2
Time Frame: Day 10 at age-specific times
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/mL/(mg/kg)
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ng*h/mL/(mg/kg)
  Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  Cannabidiol | 115.8 (55.32) | 106.0 (94.64) | 135.7 (89.17)
  7-OH Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  7-OH Cannabidiol | 102.2 (53.01) | 80.19 (63.53) | 108.7 (70.76)

23. Primary Outcome: Minimum Plasma Concentration (Cmin) for Cannabidiol and Metabolite 7-OH Cannabidiol
Description: as for outcome 2
Time Frame: Day 10 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for Cmin.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ng/mL
  Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  Cannabidiol | 19.97 (8.798) | 41.67 (25.41) | 118.3 (75.82)
  7-OH Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  7-OH Cannabidiol | 21.82 (13.23) | 34.11 (23.99) | 108.7 (70.87)

24. Primary Outcome: Average Plasma Concentration (Cavg) for Cannabidiol and Metabolite 7-OH Cannabidiol
Description: as for outcome 2
Time Frame: Day 10 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for Cavg.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ng/mL
  Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  Cannabidiol | 48.56 (23.58) | 91.38 (80.92) | 225.7 (149.3)
  7-OH Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  7-OH Cannabidiol | 42.94 (22.54) | 69.37 (56.09) | 180.4 (117.1)

25. Primary Outcome: Accumulation Ratio for Cmax (RCmax) on Day 10 for Cannabidiol and Metabolite 7-OH Cannabidiol
Description: RCmax is the ratio of Cmax at Day 10 compared to Cmax at Day 1.
  Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2 years: Day 10 pre-dose and at 2, 4, 8 and 12 hours post-dose; Participants ages 2 to <6 years: Day 10 pre-dose and at 1, 2, 3, 4, 8, 12 and 24 hours post-dose; Participants ages 6 to ≤17 years: Day 10 pre-dose and at 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
Time Frame: Day 10 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for RCmax.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ratio
  Cannabidiol: number analyzed (Participants) | 20 | 17 | 21
  Cannabidiol | 5.535 (5.551) | 4.454 (4.466) | 7.488 (11.93)
  7-OH Cannabidiol: number analyzed (Participants) | 20 | 17 | 21
  7-OH Cannabidiol | 3.823 (2.730) | 3.996 (3.544) | 5.788 (6.028)

26. Primary Outcome: Accumulation Ratio for AUC(0-12) [RAUC(0-12)] on Day 10 for Cannabidiol and Metabolite 7-OH Cannabidiol
Description: RAUC(0-12) is the ratio of AUC(0-12) at Day 10 compared to AUC(0-12) at Day 1.
  Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 1 to <2 years: Day 10 pre-dose and at 2, 4, 8 and 12 hours post-dose; Participants ages 2 to <6 years: Day 10 pre-dose and at 1, 2, 3, 4, 8, 12 and 24 hours post-dose; Participants ages 6 to ≤17 years: Day 10 pre-dose and at 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose.
Time Frame: Day 10 at age-specific times
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for RAUC(0-12).
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
ratio
  Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  Cannabidiol | 5.434 (3.625) | 5.489 (4.633) | 9.376 (15.11)
  7-OH Cannabidiol: number analyzed (Participants) | 19 | 17 | 21
  7-OH Cannabidiol | 4.865 (2.748) | 4.524 (3.338) | 7.541 (7.187)

27. Primary Outcome: Time Linearity Index for Cannabidiol and Metabolite 7-OH Cannabidiol in Participants ≥2 Years of Age
Description: Time linearity index is calculated as the ratio of AUC(0-12) on Day 10/AUC[0-inf] on Day 1.
  Serial blood sample collection times for pharmacokinetic (PK) analysis were based on the participant's age as follows:
  Participants ages 2 to <6 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24 and 48 hours post-dose; Participants ages 6 to ≤17 years: Day 1 pre-dose and at 1, 2, 3, 4, 8, 12, 16, 24, 36, 48 and 72 hours post-dose; Participants ages 1 to <2 years were not included in this analysis.
Time Frame: Day 1 and Day 10
Population: PK Population, all participants who received ≥1 dose of study drug and had ≥1 post-dose measured plasma concentration of cannabidiol and/or 7-OH cannabidiol with evaluable PK data available for analysis. The number of participants in each category is the number of participants with evaluable PK data available for time linearity index.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 15 | 15 | 16
ratio
  Cannabidiol: number analyzed (Participants) | 9 | 6 | 12
  Cannabidiol | 3.211 (2.048) | 2.628 (2.276) | 4.201 (4.990)
  7-OH Cannabidiol: number analyzed (Participants) | 14 | 9 | 13
  7-OH Cannabidiol | 2.500 (0.9365) | 1.821 (1.162) | 3.045 (2.260)

28. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product. It does not necessarily have a causal relationship with this treatment. A TEAE was defined as any event not present prior to the initiation of the treatment or any event already present that worsens. Any laboratory (clinical chemistry, hematology, urinalysis), 12-lead electrocardiograms, vital signs (temperature, blood pressure, pulse rate, respiratory rate) and physical examination findings deemed by the investigator to be clinically significant were captured as AEs. A SAE is any untoward medical occurrence that results in death, is life-threatening, requires the participant be at a risk of death at the time of the event, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect, or other serious event that requires medical or surgical intervention.
Time Frame: From the first dose of study drug up to Day 17
Population: Safety Analysis Population (SAF), all participants who received ≥1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
Participants
  TEAE | 13 | 9 | 17
  SAE | 0 | 1 | 2

29. Primary Outcome: Clinical Global Impression of Improvement (CGI-I) Assessment
Description: The CGI-I was completed by the parents/caregivers and the investigator and was used to assess participants global status of their condition on Day 11 using a 7-point scale, where 1=very much improved and 7=very much worse since the initiation of treatment.
Time Frame: Day 11
Population: Efficacy Analysis Population (EFF), all participants who received ≥1 dose of the investigational product and had ≥1 efficacy assessment for CGI-I post-dose.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
scores on a scale
  Parents/Caregivers | 2.1 (1.02) | 2.4 (0.82) | 2.3 (1.15)
  Investigator | 2.7 (0.92) | 2.5 (0.94) | 2.9 (0.91)

30. Primary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Assessment
Description: The CGI-S was completed by the parents/caregivers and the Investigator and was used to rate participant's mental illness status at Baseline (Screening) and Day 11 using a 7-point scale, where 1=normal, not mentally ill, and 7=among the most extremely mentally ill participants. This rating is based upon observed and reported symptoms, behavior, and function in the past seven days. The change in CGI-S score at Day 11 relative to Baseline is reported. A negative change from Baseline indicates improvement (decreased severity in illness).
Time Frame: Baseline and Day 11
Population: EFF, all participants who received ≥1 dose of the investigational product and had ≥1 efficacy assessment for CGI-S post-dose.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
scores on a scale
  Parents/Caregivers: number analyzed (Participants) | 17 | 19 | 21
  Parents/Caregivers | -1.7 (2.08) | -2.2 (2.04) | -1.8 (1.64)
  Investigator: number analyzed (Participants) | 17 | 19 | 21
  Investigator | -1.1 (1.27) | -0.7 (1.15) | -0.7 (1.23)

31. Primary Outcome: Change From Baseline in Daily Seizure Activity
Description: The specific number of tonic and atonic seizures per study day were recorded in a diary. The change in number of seizures at Day 11 relative to Baseline is reported. A negative change from Baseline indicates an improvement based on Daily Seizure Activity.
Time Frame: Baseline and Day 11
Population: EFF, all participants who received ≥1 dose of the investigational product and had ≥1 efficacy assessment for number of seizures per day at Day 11.
Measure: Mean (Standard Deviation); unit: number of seizures per day
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 20 | 20 | 21
number of seizures per day
  Number of Tonic Seizures: number analyzed (Participants) | 19 | 13 | 19
  Number of Tonic Seizures | -0.8 (1.55) | -0.8 (1.59) | -2.9 (7.69)
  Number of Atonic Seizures: number analyzed (Participants) | 19 | 13 | 19
  Number of Atonic Seizures | -0.2 (0.98) | -0.1 (0.28) | 0.0 (0.00)

32. Primary Outcome: Number of Participants With Suicide Related Thoughts and Behaviors Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captured the occurrence, severity, and frequency of suicide related thoughts and behaviors at Day 11. The C-SSRS was only used for participants ≥ 7 years of age. The number of participants with results of "Yes" for Suicidal Ideation (Wish to be Dead and Non-Specific Active Suicidal Thoughts) and Suicidal Behavior (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior, and Suicidal Behavior) are reported.
Time Frame: Day 11
Population: Participants from the Safety Analysis Population (SAF), all participants who received ≥1 dose of the investigational product, who completed the C-SSRS.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
Number analyzed (Participants) | 4 | 5 | 4
Participants
  Suicide Ideation | 0 | 0 | 0
  Suicide Behavior | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to 7 days after the last dose of study drug (up to Day 17)
Description: Participants who completed all study activities for this study had the option to participate in a rollover study. Participants who enrolled into the rollover study may not have had adverse event data collected after Day 11.
Arm/Group | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] | High Dose Cannabidiol Oral Solution [40 mg/kg/Day]
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20 | 2/21
Other Adverse Events (participants affected / at risk) | 13/20 | 9/20 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] (N=20) | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] (N=20) | High Dose Cannabidiol Oral Solution [40 mg/kg/Day] (N=21)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Cannabidiol Oral Solution [10 mg/kg/Day] (N=20) | Mid Dose Cannabidiol Oral Solution [20 mg/kg/Day] (N=20) | High Dose Cannabidiol Oral Solution [40 mg/kg/Day] (N=21)
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 7
Flatulence (Gastrointestinal disorders) | 0 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Catheter site pruritus (General disorders) | 0 | 2 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Somnolence (Nervous system disorders) | 3 | 3 | 7
Psychomotor hyperactivity (Nervous system disorders) | 0 | 2 | 3
Seizure (Nervous system disorders) | 1 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0
Lice infestation (Infections and infestations) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Blood follicle stimulating hormone increased (Investigations) | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Blood follicle stimulating hormone decreased (Investigations) | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1
Sedation (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Alanine aminotransferase increase (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No